CLINICAL TRIAL: NCT06624540
Title: Effect of Implementing Evidence-based Practice and Nurse's Behavior Change on Quality of Care in Intensive Care Unit: Focus on Ventilator Associated Pneumonia in a Tertiary Hospital in Bangladesh
Acronym: EBP in Nursing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Nahida Akhter, Principal Investigator, Ph.D Fellow, Graduate School of Biomedical and Health Sciences, Hiroshima University, Japan., Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BMRC/NREC/2022-2025/338; 584 19 05 2024 (Registry Identifier: BMRC (Bangladesh Medical Research Council)); 24K02733 (Registry Identifier: Japan Society for the Promotion of Science (JSPS))
Record Dates: First submitted 2024-09-12; First posted 2024-10-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Ventilator Associated Pneumonia (VAP); Evidence Based Practice
Keywords: evidence based practice; Ventilator Associated Pneumonia; Nurses Knowledge
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Phase 1: Incidence of adverse events in ICU(VAP rate, MDRPU rate, PU rate, CLABSI rate) length of stay, survival rate.
  Phase 2: A pre- and post- quasi-experimental study to evaluate the knowledge and skill of nurses.
  Phase 3: A pre- and post- quasi-experimental study to evaluate the outcomes of the patients in the ICU, using study 1 historical data as a control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Phase 2: All Nurses in GICU; Phase 3: All patients admitted in the general GICU (Experimental): Nurses: All nurses who work at GICU of DMCH Patients: all patients who will admit at the assigned GICU during the study period of DMCH
  Interventions: Behavioral: This is a pre- and post- quasi-experimental study.; Behavioral: Education with EBP

INTERVENTIONS:
Behavioral: This is a pre- and post- quasi-experimental study. — We will use new equipment and implement EBP (VAP management) for patients by trained nurses (Phase 2) and check the outcome of the patients. We will compare our phase 1 findings for this study as historical data.
Behavioral: Education with EBP — Phase 2: Nurse's EBP training ( VAP management), 2 hours lecture and 3 hours skill training for total 4 times in 1 month.
  Phase 3: Introduce new equipment necessary for EBP implementation for VAP management, and EBP-trained nurses implementation for VAP management.
  Other Names: Phase 2: Nurses EBP training

SUMMARY:
Quality of care is crucial for preventing adverse events such as infection in the intensive care units (ICUs). The most common ICU-acquired infections include pneumonia such as ventilator-associated pneumonia (VAP), Central Line Bloodstream Infection (CLABSI), catheter-associated urinary tract in, Medical Device Related Pressure Ulcer (MDRPU) and Pressure Ulcer (PU). This study explores the patient outcome in ICU by examining the causes and prevalence of ICU-acquired infection. The implementation of evidence-based practice (EBP) to reduce infection and change the nurses practice (behavioral changes) to adhere with EBP based on simulation-based training.

General objective:

To evaluate the effect of EBP by using recent technologies-based equipment to prevent VAP and promote behavior change among nurses for better outcome of the patient in ICU.

Specific Objectives:

1. To determine the incidence of adverse events (VAP rate, MDRPU rate, PU rate, CLABSI rate), length of stay and survival rate in ICU.
2. To evaluate the effectiveness of EBP education by changing nurses' behavior and determine its impact on improving patient outcomes in the ICU.
3. To evaluate the effectiveness of EBP including proper equipment use and changed nurses behavior acquired through the training for better patient outcome (VAP ratio) in the ICU.
4. To examine the feasibility of evaluation process and outcomes and successful implementation of EBP in ICU.

Hypothesis:

It is hypothesize that implementing EBP in ICU, including new equipment use and nurses training, will improve patient outcome.

These research consist of three studies:

Phase 1: Incidence of adverse events (VAP rate, MDRPU rate, PU rate, CLABSI rate), length of stay and survival rate in ICU. The patients of General ICU will be followed up after admission up to discharge or death at ICU. The investigators use the study findings for our subsequent intervention study 3 as historical data.

Phase 2: A pre- and post- quasi-experimental study will be conducted for 6 months to evaluate the nurse's competency on EBP after getting 1-month EBP training. This study has 3 steps: (1) Pre-observation period to measure nurse's competency level for 2-month, (2) nurse's EBP training period with preparation for 1 month, and (3) post-implementation period to measure nurse's competency and implementation of EBP practice for 2 months. Study nurses will receive EBP training, EBP and proper equipment for patient management. The nurses will receive EBP education and training with necessary equipment, such as a close suction catheter, an endotracheal tube, a suction device, and a mouth care brush. In this study, use global standard equipment for the patients safety.

Phase 3: A pre- and post- quasi-experimental study will be implemented to evaluate the efficacy of EBP implementation. The investigators use new equipment and implement EBP for patients and assess the patient outcomes. The investigators compare the findings from study 1 (as historical data) with the data from this study 3.

The investigators will compare the VAP infection prevalence and patients' outcomes related to ICU-acquired infection between pre- and post- test phase.

ELIGIBILITY:
Study 2:

Inclusion criteria:

* Who will be a registered nurse in Bangladesh.
* Who will agree to participate in this study and the EBP training.

Exclusion criteria:

* Who will not directly involve patient care in ICU.

Study 3:

Inclusion Criteria:

* Irrespective of age and sex, participant must be 18 years old.
* Legal guardian of a patient consents to participation in the study
* Intubated patients after admission.

Exclusion Criteria:

* Who stays less than 2 days at the GICU.
* Who dies or is extubated within 2 days after admitted in the GICU.
* ICU readmission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The nurse's skill performance is related to VAP checklist | Study 2: 6 months
  Nurses' skill performance related to VAP prevention measured using a researcher-developed 64-item observational checklist based on evidence-based practice guidelines.
  Unit of Measure: Total skill performance score (range 0-140), categorized as:
  * High: ≥112 (≥80%)
  * Moderate: 70-111 (50-79%)
  * Low: <70 (<50%)
Incidence rate of ventilator-associated pneumonia (VAP) | 2 months
  Number of new ventilator-associated pneumonia cases occurring in ICU patients during the study period. Unit of Measure: VAP cases per 1,000 ventilator days.
  Data will be collected: Patients' demographic data (age, sex, occupation etc.) Medical past and current history (diagnosis, treatment, medication, hospitalization). Reasons and date to be admitted to ICU. Treatment in ICU. Daily laboratory data taken in ICU. Daily biological data including vital signs. Results of patients' stay during ICU. Duration of ventilation Diagnosis of VAP

SECONDARY OUTCOMES:
A nurse's motivation level will be measured | 6 month
  A nurse's motivation level will be measured by the Motivation scale. . Total 12 items, and score ranges 1 lower motivation and 10 higher motivations.
Nurses' sustained implementation measured | 6 months
  Nurses' sustained implementation measured by Nurses sustained implementation scale. The total item is 28, and 4-point liker scale. Scores ranges from 28 (no sustainability) to 112 (good sustainability).
Organizational readiness measured | 6 months
  Organizational readiness measured by Organizational readiness scale. Total 03 items convergent validity (r = 0.42 - 0.72) for the correlations between the shortened and longer scales.
Nurses knowledge and practice related to VAP prevention measured. | 6 months
  Measured by researcher modified nurses knowledge related to VAP prevention scale total 12 & 6 items.
VAP episode | 2 months
  Number of new ventilator-associated pneumonia cases occurring in ICU patients during the study period.
Interval of VAP occurrence | 2 months
  Number of days from date/time of ICU admission to date/time of first diagnosis of ventilator-associated pneumonia (VAP). If no VAP occurs, observation is censored at ICU discharge or death.
  Unit of Measure: Days (time-to-event) - report as median (IQR) and mean ± SD; consider Kaplan-Meier estimates for time-to-event.
Micro-organism link to VAP | 2 months
  After diagnosis of CLABSI then identify what kind organism relate to CLABSI. Type and frequency of microorganisms identified in laboratory-confirmed CLABSI cases. Unit of Measure: Number of cases per microorganism
Mortality and morbidity rate | 2 months
  Mortality and morbidity rate of ICU patients All-cause mortality among ICU patients during the study period. Unit of Measure: Percentage (%)。Occurrence of ICU-related adverse events (VAP). Unit of Measure: Number of patients with adverse events
Onset of VAP | 2 months
  Classification of first VAP episode as early-onset or late-onset based on time from initiation of mechanical ventilation.
  Unit of Measure: Number and percentage (%) of patients with early-onset and late-onset VAP.
Length of stay ICU patients | 2 months
  Average length of stay ICU patients. Mean length of stay in the intensive care unit for enrolled patients. Unit of Measure: Days (mean ± SD)
Survival rate in ICU | 2 months
  Average survival rate of ICU. Data will be collected: Length of stay and survival rate. Proportion of enrolled patients alive at ICU discharge. Unit of Measure: Percentage (%) of patients surviving to ICU discharge.

CONTACTS AND LOCATIONS:
Locations (2):
- Dhaka Medical College Hospital, Dhaka, Bangladesh
- Hiroshima University, Hiroshima, Kasumi 1-2-3 Minami-ku, Japan

IPD SHARING:
Plan to Share IPD: No
IPD will not be share due to personal confidentiality of the participants. When the data will be available and we will share the data according to the recommendations of the clinical trial registration and the requests of the journals.

REFERENCES:
- [Derived] Akhter N, Zhou X, Elhabashy S, Huq KATME, Okamoto M, Latif MA, Babaita AO, Moriyama M. Effect of evidence-based education program with mentoring system for prevention of ventilator-associated pneumonia on nurses' competency to improve quality care for patients in the intensive care unit: a quasi-experimental study in a tertiary hospital in Bangladesh. Front Public Health. 2026 Jan 9;13:1674223. doi: 10.3389/fpubh.2025.1674223. eCollection 2025. PMID 41584199